CLINICAL TRIAL: NCT00470353
Title: A Pilot Study of Low and High Dose Vitamin Cholecalciferol (D3) With Pharmacokinetic and Pharmacodynamic Correlates in Patients With Resected Colon Cancer
Brief Title: Cholecalciferol and Calcium Carbonate in Treating Patients With Colon Cancer That Has Been Removed by Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to poor accrual/lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: I 78706; RPCI-I-78706
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Calcium Carbonate; Cholecalciferol; Immunohistochemistry; Biopsy

INTERVENTIONS:
Dietary Supplement: calcium carbonate
Dietary Supplement: cholecalciferol
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: biopsy

SUMMARY:
RATIONALE: The use of cholecalciferol and calcium carbonate may keep colon cancer from coming back in patients with colon cancer that has been removed by surgery.

PURPOSE: This randomized clinical trial is studying two different doses of cholecalciferol to compare how well they work when given together with calcium carbonate in treating patients with colon cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the antiproliferative effects of 2 different doses of cholecalciferol (i.e., vitamin D3) in combination with calcium carbonate on the proliferative labeling index in patients with resected colon cancer.

Secondary

* Compare the effects of these doses on serum levels of 25-OH-D3, 1,25-OH-D3, 24,25-OH-D3, calcium, and parathyroid hormone in these patients.
* Determine the safety of high-dose cholecalciferol in these patients over 2 years.
* Compare the effects of these doses on several biological markers (i.e., cyclin D1, protein kinase C, vitamin D receptor, p21, and p27) in the rectal mucosa of these patients.

OUTLINE: This is a randomized, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral low-dose cholecalciferol once daily and oral calcium carbonate twice daily.
* Arm II: Patients receive oral high-dose cholecalciferol once daily and calcium carbonate as in arm I.

Treatment in both arms continues for up to 2 years in the absence of disease progression or unacceptable toxicity. All patients undergo sigmoidoscopy or colonoscopy with 4 quadrant mucosal biopsies at baseline and after 6 months of study treatment. After their 6-month mucosal biopsy, patients in arm I switch to high-dose cholecalciferol as in arm II.

Patients undergo blood, urine, and tissue collection periodically during study for pharmacokinetic, pharmacodynamic, and/or histopathological analysis. Serum is collected monthly for 3 months and then once every 3 months to assess changes in serum levels of vitamin D and vitamin D metabolites (i.e., 1,25-OH-D3; 25-OH-D3; 24,25-OH-D3), as well as changes in calcium and parathyroid hormone, BUN, creatinine, electrolytes, and phosphorus levels. Urine is collected once every 3 months to assess changes in urine calcium and creatinine levels for hypercalciuria. Tissue biopsies of normal endorectal mucosa collected at baseline and after 6 months of study treatment are evaluated by IHC for proliferative index, vitamin D receptor staining, p21, p27, cyclin D1, and protein kinase C.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of colon cancer

  * Underwent resection and has been in clinical remission for ≥ 1 year
* No inflammatory bowel disease
* No familial adenomatous polyposis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 1 year
* No genitourinary stones within the past 5 years
* No severe comorbid conditions, such as uncompensated heart failure or active uncontrolled infection
* No history of hypercalcemia
* No active colostomy
* No contraindications to sigmoidoscopy or mucosal biopsies

PRIOR CONCURRENT THERAPY:

* No prior rectal surgery or abdominoperineal resection
* At least 1 month since prior vitamin D or calcium supplementation

  * Prior vitamin D supplemental intake ≤ 800 IU per day
* At least 1 year since prior chemotherapy
* No prior radiotherapy to the pelvis
* No concurrent active anticoagulation

  * Patients who stop anticoagulation therapy at the time of mucosal biopsy are eligible
* No other concurrent supplemental calcium or vitamin D

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-09; Primary Completion 2008-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in proliferative labeling index of normal rectal mucosa as measured by Ki67 IHC staining

SECONDARY OUTCOMES:
Changes in serum levels of 25-OH-D3, 1,25-OH-D3, 24,25-OH-D3, calcium, and parathyroid hormone
Safety of high-dose cholecalciferol supplementation as measured over 2 years | over 2 years
Effects of cholecalciferol on biological markers of proliferation (i.e., cyclin D1, protein kinase C, vitamin D receptor, p21, and p27) as measured by IHC at baseline and after 6 months of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States